CLINICAL TRIAL: NCT03117504
Title: Assessment of Prevalence of Stress Urinary Incontinence During Pregnancy
Status: Suspended | Type: Observational
Why Stopped: lack of funding
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohammed Nour Allah Abdel Monem, Resident of obstetrics&gynecology, Ain Shams Maternity Hospital
Other Study IDs: MNAAMonem
Record Dates: First submitted 2017-03-21; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First trimester: women during first trimester(less than 14 weeks of pregnancy) will complete self-reported questionnaires and undergo clinical examination to confirm the stress incontinence.
  Interventions: Other: questionnaire
- Third trimester: women during third trimester(more than 28 weeks of pregnancy) will complete self-reported questionnaires and undergo clinical examination to confirm the stress incontinence.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — a questionnaire is given to each woman to determine the urinary incontinence and it's impact on quality of life.

SUMMARY:
Stress urinary incontinence is the most common type of incontinence during pregnancy.our study aims at determining the prevalence in the first and third trimesters and the associated risk factors.

DETAILED DESCRIPTION:
The required sample size has been calculated using IBM© Sample Power© version 3 .The primary outcome measure is the prevalence of stress urinary incontinence (SUI) in the 1st and 3rd trimesters.

Accordingly, it is estimated that a sample of 240 patients in either study group would have a power of 80% (beta error, 0.2) to detect a statistically significant difference of 9% between the two groups as regards the incidence of SUI.

The incidence of SUI is assumed to equal 10% in the 1st trimester. The prevalence of SUI in the 3rd trimester is assumed to equal 10% under the null hypothesis and to equal 19% under the alternative hypothesis.

This calculation used a two-sided z test with a confidence level of 95% (alpha error, 0.05).

Data will be collected, tabulated, then analyzed using IBM© SPSS© Statistics version 22.

Normally distributed numerical data will be presented as mean and SD, and skewed data as median and inter-quartile range.

Qualitative data will be presented as number and percentage.Comparison of normally distributed numerical data will be done using the unpaired Student t test. Skewed data will be compared using the Mann-Whitney U test.

Categorical data will be compared using the chi-squared test, or Fisher's exact test when appropriate.

A two-sided p-value <0.05 will be considered statistically significant .

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in first and third trimesters

Exclusion Criteria:

* Communication problems.
* Mental disturbances.
* Previous surgery for incontinence or other pelvic procedures.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: A cross-sectional study of two groups of women will be conducted. Each group consists of 250 patients with a total number of 500 patients
  * group 1 : women during first trimester(less than 14 weeks of pregnancy).
  * group 2: women during third trimester (more than 28 weeks of pregnancy).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-05-20 (Estimated); Study Completion 2017-07-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stress urinary incontinence during first trimester pregnancy | 2 years
  Determine the prevalence and associated risk factors in the first trimester

SECONDARY OUTCOMES:
Prevalence of stress urinary incontinence during third trimester pregnancy | 2 years
  Determine the prevalence and associated risk factors in the third trimester

CONTACTS AND LOCATIONS:
Overall Officials: Hazem M Sammour, MD, Study Chair — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Faculty of Medicine, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No